CLINICAL TRIAL: NCT02551874
Title: A 24-week International, Multicenter, Randomized, Open-Label, Active-Controlled, Parallel Group, Phase 3b Trial With a 28-week Extension to Evaluate the Efficacy and Safety of Saxagliptin Co-administered With Dapagliflozin Compared to Insulin Glargine in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin With or Without Sulfonylurea Therapy
Brief Title: A 24-week Open-Label, Phase 3b Trial With a 28-week Extension to Evaluate the Efficacy and Safety of Saxagliptin Co-administered With Dapagliflozin Compared to Insulin Glargine in Subjects withType 2 Diabetes Who Have Glycemic Control on Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV181-369; 2015-001702-33 (EudraCT Number)
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; dapagliflozin; Insulin Glargine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin/Dapagliflozin/Metformin (Experimental): Oral route. Saxagliptin/Dapa adminsitered once daily for 24 weeks at a dose of 5 mg Saxagliptin and 10 mg Dapagliflozin
  Interventions: Drug: Saxagliptin, Onglyza; Drug: Dapagliflozin, Farxiga; Drug: Metformin
- Insulin Glargine, Lantos/Metformin (Active Comparator): Insulin glargine administered once a day with starting dose of 0.2 Unit per kg or 10 units.
  Interventions: Drug: Glargine insulin

INTERVENTIONS:
Drug: Saxagliptin, Onglyza — Tablets, Oral, 5mg , Once daily, 24 weeks
  Other Names: Onglyza
  Arms: Saxagliptin/Dapagliflozin/Metformin
Drug: Dapagliflozin, Farxiga — Tablets, Oral, 10mg , Once daily, 24 weeks
  Other Names: BMS-512148
  Arms: Saxagliptin/Dapagliflozin/Metformin
Drug: Glargine insulin — 100 Units/ml solution for injection in a prefilled SoloStar pen
  Other Names: Lantus
  Arms: Insulin Glargine, Lantos/Metformin
Drug: Metformin — Tablets, Oral, ≥ 1500mg/≤ 2500mg, Once daily, 24 weeks
  Other Names: Glucophage
  Arms: Saxagliptin/Dapagliflozin/Metformin

SUMMARY:
This research study of subjects with inadequately controlled type 2 diabetes mellitus (T2DM) will compare the glycemic control (measured by HbA1c) in subjects co-administered saxagliptin and dapagliflozin, in addition to metformin with or without sulfonylurea, to subjects receiving insulin glargine, in addition to metformin with or without sulfonylurea, over a treatment period of 52 weeks.

DETAILED DESCRIPTION:
CV181-369; A 24 Week International, Open-Label Trial With a 28 Week Extension to Evaluate the Efficacy of Saxagliptin Co-administered With Dapagliflozin Compared to Insulin Glargine in Subjects With Type 2 Diabetes on Metformin With or Without Sulfonylurea Therapy

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* At least 18 years of age at screening
* HbA1c ≥ 8% and ≤ 12% at screening
* Fasting plasma glucose (FPG) ≤ 270 mg/dL (15mmol/L)
* Stable dose metformin ≥ 1500 mg per day with or without a stable dose of sulfonylurea (defined as at least 50% maximal dose per local label) for at least 8 weeks
* estimated glomerular filtration rate (eGFR) < 60 ml/ml/1.73m2
* Body Mass Index ≤ 45.0 kg/m2

Exclusion Criteria:

* Clinical diagnosis of Type 1 diabetes
* History of ketoacidosis
* Renal, hepatic or pancreatic disease
* Impairment of renal function (defined as creatinine clearance [CrCl] < 60 mL/min
* Cardiovascular or vascular diseases identified within 3 months of participationImpairment of renal function (defined as creatinine clearance [CrCl] < 60 mL/min

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca, Study Director — AstraZeneca
Locations (35):
- United States (18):
  - Research Site, Anaheim, California
  - Research Site, Los Angeles, California
  - Research Site, Miami, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Norcross, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Quincy, Massachusetts
  - Research Site, Beavercreek, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Barto, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Bountiful, Utah
- Czechia (2):
  - Research Site, Karlovy Vary
  - Research Site, Olomouc
- Research Site, Copenhagen, Denmark
- Research Site, Budapest, Hungary
- Mexico (4):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Zapopan, Jalisco
- Poland (3):
  - Research Site, Lodz
  - Research Site, Nowy Duninów
  - Research Site, Sochaczew
- Romania (3):
  - Research Site, Craiova
  - Research Site, Ploieşti
  - Research Site, Timișoara
- Research Site, Lenasia, South Africa
- Research Site, A Coruña, Spain
- Research Site, Uddevalla, Sweden

REFERENCES:
- [Derived] Vilsboll T, Ekholm E, Johnsson E, Dronamraju N, Jabbour S, Lind M. Dapagliflozin Plus Saxagliptin Add-on Therapy Compared With Insulin in Patients With Type 2 Diabetes Poorly Controlled by Metformin With or Without Sulfonylurea Therapy: A Randomized Clinical Trial. Diabetes Care. 2019 Aug;42(8):1464-1472. doi: 10.2337/dc18-1988. Epub 2019 Jun 4. PMID 31167892
- See also: cv181-369 SAP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4129&filename=cv181-369_SAP_redacted.pdf
- See also: cv181-369 CSP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4129&filename=cv181-369_CSP_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 112 centers in 11 countries from 20 Oct 2015 to 10 Nov 2017. There were 2 data cut-offs for this study: 8 May 2017 for analyses of the short-term study period (after 24 weeks of open-label treatment) and 10 Nov 2017 for analyses of the short-term plus long-term study period (after 52 weeks of open-label treatment).
Pre-assignment Details: The study duration was up to 56 weeks, consisting of a 2-week screening period, 2-week lead-in period, 24-week short-term treatment period, and 28-week long-term treatment period.
Groups:
- Dapagliflozin + Saxagliptin + Metformin: Subjects received dapagliflozin 10 milligrams (mg) and saxagliptin 5 mg, administered orally once daily (QD) in the morning for the 52-week treatment period (24-week short-term period and 28-week long term period).
  Subjects continued to receive their stable dose of metformin with or without sulfonylurea (SU) throughout the study.
- Titrated Insulin + Metformin: Subjects were to administer insulin glargine subcutaneously QD at the same time every day for the 52-week treatment period (24-week short-term period and 28-week long term period), following investigator instructions and training. All subjects started with an initial dose of 0.2 units/kilogram (kg) body weight or at least 10 units of insulin per day. Subjects self-titrated the dose of insulin glargine over the first 8 weeks of the study based on daily glucose monitoring. The investigator had the discretion to modify insulin dose based on his/her assessment between Week 8 and Week 12 with the goal to reach an acceptable and stable insulin dose by Week 12.
  Subjects continued to receive their stable dose of metformin with or without SU throughout the study.
Period: Overall Study
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Titrated Insulin + Metformin
Started | 324 | 326
Received Treatment in Short-term Study | 324 | 319
Entered Long-term Study | 306 | 294
Received Treatment in Long-term Study | 295 | 284
Completed | 296 | 287
Not Completed | 28 | 39
Not completed — Lost to Follow-up | 0 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Reason not reported | 10 | 4
Not completed — Did not receive randomized treatment | 0 | 7
Not completed — Did not enter long-term study | 18 | 25

BASELINE CHARACTERISTICS:
Groups:
- Dapagliflozin + Saxagliptin + Metformin: Subjects received dapagliflozin 10 mg and saxagliptin 5 mg, administered orally QD in the morning for the 52-week treatment period (24-week short-term period and 28-week long term period).
  Subjects continued to receive their stable dose of metformin with or without SU throughout the study.
- Titrated Insulin + Metformin: Subjects were to administer insulin glargine subcutaneously QD at the same time every day for the 52-week treatment period (24-week short-term period and 28-week long term period), following investigator instructions and training. All subjects started with an initial dose of 0.2 units/kg body weight or at least 10 units of insulin per day. Subjects self-titrated the dose of insulin glargine over the first 8 weeks of the study based on daily glucose monitoring. The investigator had the discretion to modify insulin dose based on his/her assessment between Week 8 and Week 12 with the goal to reach an acceptable and stable insulin dose by Week 12.
  Subjects continued to receive their stable dose of metformin with or without SU throughout the study.
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Titrated Insulin + Metformin | Total
Number analyzed (Participants) | 324 | 319 | 643
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (9.52) | 55.3 (9.63) | 55.5 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 148 | 296
  Male | 176 | 171 | 347
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 12 | 6 | 18
  Asian | 12 | 12 | 24
  Black Or African American | 28 | 35 | 63
  Native Hawaiian Or Other Pacific Islander | 0 | 1 | 1
  Other | 9 | 11 | 20
  White | 263 | 254 | 517

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in HbA1c at Week 24
Description: To examine whether the mean change from baseline in HbA1c with co-administered saxagliptin 5 mg and dapagliflozin 10 mg plus metformin with or without SU is noninferior (noninferiority margin of 0.3%) to titrated insulin glargine plus metformin with or without SU after 24 weeks of open-label treatment.
Time Frame: Baseline and Week 24
Population: The randomized subjects data set consisted of all randomized subjects who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: % HbA1c
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Titrated Insulin + Metformin
Number analyzed (Participants) | 319 | 312
% HbA1c | -1.67 [-1.79 to -1.55] | -1.54 [-1.66 to -1.42]
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Titrated Insulin + Metformin; Test type: Non-Inferiority — Noninferiority was defined by upper bound of 95% CI <0.3%; p = 0.118, Mixed Models Analysis — Superiority; Adjusted for treatment, baseline HbA1c, randomization stratification factor, visit, treatment-by-visit, and baseline HbA1c-by-visit; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.30 to 0.03], Standard Error of Mean 0.085

2. Secondary Outcome: Mean Change From Baseline in Total Body Weight at Week 24
Description: To compare the mean change from baseline in total body weight with co-administered saxagliptin 5 mg and dapagliflozin 10 mg plus metformin with or without SU versus titrated insulin glargine plus metformin with or without SU after 24 weeks of open-label treatment
Time Frame: Baseline and Week 24
Population: The number of participants is the number of subjects in the randomized subject data set with non-missing baseline assessments and at least one post-baseline assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Titrated Insulin + Metformin
Number analyzed (Participants) | 319 | 313
kg | -1.50 [-1.89 to -1.11] | 2.14 [1.75 to 2.54]
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Titrated Insulin + Metformin; Test type: Superiority; p < 0.001, Mixed Models Analysis; Adjusted for treatment, baseline body weight, randomization stratification factor, visit, treatment-by-visit, and baseline body weight-by-visit; Mean Difference (Final Values) = -3.64, 95% CI 2-sided [-4.20 to -3.09], Standard Error of Mean 0.282

3. Secondary Outcome: Percentage of Subjects With Confirmed Hypoglycaemia at Week 24
Description: Hypoglycemia defined as plasma glucose ≤70 mg/dL (3.9 mmol/L)
Time Frame: Baseline and Week 24
Population: The randomized subject data set consisted of all randomized subjects who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Adjusted % Participants
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Titrated Insulin + Metformin
Number analyzed (Participants) | 324 | 319
Adjusted % Participants | 21.3 [17.03 to 26.22] | 38.4 [32.94 to 44.07]
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Titrated Insulin + Metformin; Test type: Superiority; p < 0.001, Regression, Logistic; Adjusted for baseline HbA1c and randomization stratification factor (background medication of metformin with or without SU); Odds Ratio (OR) = 0.4, 95% CI 2-sided [0.30 to 0.62]

4. Secondary Outcome: Percentage of Subjects Achieving a Therapeutic Glycemic Response, Without Hypoglycaemia, at Week 24
Description: To compare the percentage of subjects achieving a therapeutic glycemic response, defined as HbA1c <7.0%, without any reported hypoglycemia, with co-administered saxagliptin 5 mg and dapagliflozin 10 mg plus metformin with or without SU versus titrated insulin glargine plus metformin with or without SU after 24 weeks of open-label treatment.
Time Frame: Baseline and Week 24
Population: The randomized subject data set consisted of all randomized subjects who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Adjusted % Participants
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Titrated Insulin + Metformin
Number analyzed (Participants) | 324 | 319
Adjusted % Participants | 20.9 [16.69 to 25.83] | 13.1 [9.72 to 17.33]
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Titrated Insulin + Metformin; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.16 to 2.67]

5. Secondary Outcome: Percentage of Subjects Achieving a Therapeutic Glycemic Response at Week 24
Description: To examine whether the percentage of subjects achieving a therapeutic glycemic response, defined as HbA1c <7.0%, with co-administered saxagliptin 5 mg and dapagliflozin 10 mg plus metformin with or without SU is noninferior (noninferiority margin of 10%) to titrated insulin glargine plus metformin with or without SU after 24 weeks of open-label treatment.
Time Frame: Baseline and Week 24
Population: The randomized subject data set consisted of all randomized subjects who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Adjusted % Participants
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Titrated Insulin + Metformin
Number analyzed (Participants) | 324 | 319
Adjusted % Participants | 33.2 [28.00 to 38.79] | 33.5 [28.28 to 39.26]
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Titrated Insulin + Metformin; Test type: Non-Inferiority — Noninferiority was defined by lower bound of 95% CI >-10%; Adjusted Percent Difference = -0.4, 95% CI 2-sided [-7.42 to 6.54]

6. Secondary Outcome: Change From Baseline in the Mean Value of 24-hour Glucose at Week 2
Description: Change from baseline in the mean value of 24-hour glucose readings measured by Continuous Glucose Monitoring with co-administered saxagliptin 5 mg and dapagliflozin 10 mg plus metformin with or without SU is noninferior to titrated insulin glargine plus metformin with or without SU after 2 weeks of open-label treatment.
Time Frame: Baseline and Week 2
Population: The randomized subject data set consisted of all randomized subjects who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/deciliter (dL)
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Titrated Insulin + Metformin
Number analyzed (Participants) | 133 | 133
mg/deciliter (dL) | -48.53 [-53.47 to -43.59] | -28.54 [-33.47 to -23.61]
Statistical Analysis 1: Comparison: Dapagliflozin + Saxagliptin + Metformin vs Titrated Insulin + Metformin; Test type: Non-Inferiority — Noninferiority was defined by upper bound of 95% CI <12 mg/dL; p < 0.0001, Mixed Models Analysis; Adjusted for treatment, baseline measurement, randomization stratification factor, visit, treatment-by-visit, and baseline-by-visit; Mean Difference (Final Values) = -19.99, 95% CI 2-sided [-26.98 to -13.00], Standard Error of Mean 3.55

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) up to Week 52 (24-week short-term treatment period + 28-week long-term treatment period).
Description: Adverse event (AE) data is reported for the treated subject data set, and included AEs with an onset date on or after the date of first dose of short-term study treatment and up to and including 30 days following the date of last dose of short-term + long-term study treatment.
Arm/Group | Dapagliflozin + Saxagliptin + Metformin | Titrated Insulin + Metformin
All-Cause Mortality (participants affected / at risk) | 2/324 | 0/319
Serious Adverse Events (participants affected / at risk) | 20/324 | 13/319
Other Adverse Events (participants affected / at risk) | 55/324 | 73/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin + Saxagliptin + Metformin (N=324) | Titrated Insulin + Metformin (N=319)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Femoral hernia incarcerated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Lisfranc fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin + Saxagliptin + Metformin (N=324) | Titrated Insulin + Metformin (N=319)
Upper respiratory tract infection (Infections and infestations) | 17 (24) | 23 (26)
Viral upper respiratory tract infection (Infections and infestations) | 25 (28) | 19 (24)
Headache (Nervous system disorders) | 12 (15) | 22 (24)
Influenza (Infections and infestations) | 8 (8) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT02551874/SAP_000.pdf
  • Study Protocol (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT02551874/Prot_001.pdf